CLINICAL TRIAL: NCT06769633
Title: A Phase 2 Open-label (Core Phase Plus Extension Phase) With 2 Cohorts Study to Assess the Pharmacokinetics and Safety of Givinostat in DMD Patients Ages From at Least 2 Years to Less Than 6 Years Old
Brief Title: Pharmacokinetics and Safety of Givinostat in DMD Patients Ages From at Least 2 Years to Less Then 6 Years Old
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DSC/14/2357/52
Record Dates: First submitted 2024-12-11; First posted 2025-01-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Givinostat
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — givinostat hydrochloride; KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - from 4 to 6 years old (Experimental): Drug: Givinostat Givinostat has to be administered twice daily in a fed state according to a flexible dose regimen based on patient weight. Starting dose could be reduced based on predefined safety rules.
  Other Names:
  - ITF2357
  Interventions: Drug: Givinostat Hydrochloride
- Cohort 2 - from 2 to 4 years old (Experimental): Drug: Givinostat Givinostat has to be administered twice daily in a fed state according to a flexible dose regimen based on patient weight. Starting dose will be confirmed/adjusted with results of the interim analysis of cohort 1.
  Other Names:
  - ITF2357
  Interventions: Drug: Givinostat Hydrochloride - Cohort 2

INTERVENTIONS:
Drug: Givinostat Hydrochloride — Cohort 1 - from 4 to 6 years old
  Other Names: Cohort 1
  Arms: Cohort 1 - from 4 to 6 years old
Drug: Givinostat Hydrochloride - Cohort 2 — Cohort 2 - from 2 to 4 years old
  Other Names: Cohort 2
  Arms: Cohort 2 - from 2 to 4 years old

SUMMARY:
This is a Phase 2 Open-label (Core Phase Plus Extension Phase) With 2 Cohorts Study to Assess the Pharmacokinetics and Safety of Givinostat in younger DMD Patients.

* Planned screening duration: approximately 4 weeks
* Planned Core Treatment duration: approximately 48 weeks
* Planned Extension Treatment duration: approximately 96 weeks
* Planned Follow Up duration: approximately 4 weeks (± 7 days)
* Total duration of study participation: up to 151 weeks (ie, 37-38 months)

DETAILED DESCRIPTION:
This is an open-label, multicentre, multicountry, 2 cohorts study to evaluate the PK profile and safety of givinostat in subjects with DMD aged ≥4 to <6 years for Cohort 1 and aged ≥2 to <4 years for Cohort 2. The starting dose for Cohort 2 will be confirmed/adjusted with results of the interim analysis of Cohort 1. The study will consist of 2 phases, a Core Phase and an Extension Phase. Two final analyses will be conducted, the first at the end of the Core Phase and the second at the end of the Extension Phase (core and extension data will be combined).

The study will enrol approximately 18 subjects (approximately 9 subjects [aged ≥4 to <6 years] in Cohort 1 and approximately 9 subjects [aged ≥2 to <4 years] in Cohort 2).

ELIGIBILITY:
Inclusion Criteria - Core Phase:

1. Male children aged ≥2 to <6 years at screening (subjects ≥6 years of age at screening will not be enrolled into the study)
2. Written consent provided by parent/legal guardian and subject written assent, if applicable (according to local regulation)
3. A genetic diagnosis of DMD
4. Corticosteroid treatment considerations:

   1. For subject receiving a stable dose or oral systemic corticosteroids:

      No significant change in dose or dosing regimen (except for adjustments due to body weight change) for a minimum of 3 months immediately prior to the start of the study drug or
   2. For subjects without current corticosteroid treatment:

Must not start corticosteroids in the Core Phase of the study (ie, first 48 weeks).

Inclusion Criteria - Extension Phase:

1. Must have participated in the Core Phase study (48 weeks) and have attended the End of Treatment Visit
2. Give informed consent and /or assent in writing signed by the parent/legal guardian and/or subject (according to local regulation)
3. In stable oral systemic corticosteroids treatment with no significant change in dose or dosing regimen (except for adjustments due to body weight change). For subjects without corticosteroids during the Core Phase, the treatment can be started based on the Investigator's clinical medical judgement.

Exclusion Criteria - Core Phase

1. Exposure to another investigational drug within 3 months prior to the start of the study drug
2. Exposure to any dystrophin restoration product (eg, Ataluren, Exon skipping) within 6 months prior to the start of study drug
3. Received any gene therapy (eg, AAV Micro-dystrophin delivery) within 12 months prior to start of study drug
4. Use of any pharmacologic treatment, other than corticosteroids, that might have had an effect on muscle strength or function within 3 months prior to the start of the study drug (eg, growth hormone). Note: Vitamin D, calcium, and any other supplements will be allowed.
5. Have had surgery that might have an effect on muscle strength or function within 3 months prior to start of the study drug or planned surgery at any time during the study
6. The presence of other clinically significant disease, which, in the Investigator's opinion, could adversely affect subject's safety, making it unlikely to complete the study or to be compliant with study-specific requirements that could impair the assessment of study results
7. Diagnosis of other uncontrolled neurological diseases or presence of relevant uncontrolled somatic disorders that are not related to DMD, based on Investigator clinical medical judgement
8. Platelet count, white blood cells, and/or haemoglobin counts < lower limit of normal (LLN) at screening (Note: for abnormal screening laboratory test results [<LLN], the platelet count, white blood cell, and haemoglobin will be repeated once; if the repeat test result is still <LLN, the subject will be excluded)
9. Current or history of liver disease or impairment, including but not limited to a baseline elevated total bilirubin (ie, >1.5 × upper limit of normal [ULN]), unless secondary to Gilbert disease or pattern consistent with Gilbert disease
10. Inadequate renal function, as defined by serum Cystatin C result >2 × ULN (Note: if the value is >2 × ULN, the serum Cystatin C will be repeated once; if the repeated test result is still >2 × ULN, the subject will be excluded)
11. Fasting triglycerides >300 mg/dL (3.42 mmol/L) at screening (Note: if the value is >300 mg/dL, the triglycerides will be repeated once; if the repeated test result is still >300 mg/dL in fasting, the subject should be excluded)
12. Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus at screening
13. Baseline corrected QT interval using Fridericia's formula (QTcF) >450 msec (as the mean of 3 consecutive readings taken 5 minutes apart) or history of additional risk factors for torsades de pointes (ie, heart failure, hypokalaemia, or family history of long QT syndrome)
14. Psychiatric illness or social situations rendering the potential subject unable to understand and comply with the muscle function tests and/or with the study protocol procedures, based on the Investigator's clinical medical judgement
15. Hypersensitivity to any component of study drug
16. Sorbitol intolerance or malabsorption or have the hereditary form of fructose intolerance.
17. Body weight <10 kg at screening.

Exclusion Criteria - Extension Phase

1. Platelet count, white blood cells, and/or haemoglobin <LLN at EOT/V12 (Note: for abnormal laboratory test results [<LLN], the platelet count, white blood cell, and haemoglobin will be repeated once; if the repeat test result is still <LLN, the subject will be excluded)
2. Current liver disease or impairment, including but not limited to an elevated total bilirubin (ie, >1.5 × ULN), unless secondary to Gilbert disease or pattern consistent with Gilbert disease
3. Inadequate renal function, as defined by serum Cystatin C result >2 × ULN (Note: if the value is >2 × ULN, the serum Cystatin C will be repeated once; if the repeated test result is still >2 × ULN, the subject will be excluded)
4. Fasting triglycerides >300 mg/dL (3.42 mmol/L; Note: if the value is >300 mg/dL, the triglycerides will be repeated once; if the repeated test result is still >300 mg/dL in fasting condition, the subject should be excluded)
5. Have presence of other clinically significant disease, which, in the Investigator's opinion, could adversely affect the safety of the subject, making it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results
6. Evidence of psychiatric illness or social situations rendering the potential subject unable to understand and comply with the muscle function tests and/or with the study protocol procedures, based on the Investigator's clinical medical judgement.

Ages: 2 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Core Phase: Cohort 1 - Change from baseline of the pharmacokinetic (PK) parameter Area under the concentration-time curve from dosing (time 0) to time t at steady state (AUC0-T,ss). | Baseline up to week 48
  Pharmacokinetic samples will be collected 1 pre-dose in the morning and 3 post-dose (0-2 h, 4-6 h, 6-8 h) after 1 week (Visit 3) and after 6 months (Visit 10). Sampling times will be randomly assigned to each subject to collect at least 1 pre-dose sample and 2 post-dose samples in each subject. At these timepoints, the subject will be asked to take the morning dose at the site. Samples collected after 1 week of treatment will be used for the exploratory PK analysis.
Core Phase: Cohort 1 - Change from baseline of the pharmacokinetic (PK) parameter maximum plasma concentration at steady state (Cmax,ss). | Baseline up to week 48
  Pharmacokinetic samples will be collected 1 pre-dose in the morning and 3 post-dose (0-2 h, 4-6 h, 6-8 h) after 1 week (Visit 3) and after 6 months (Visit 10). Sampling times will be randomly assigned to each subject to collect at least 1 pre-dose sample and 2 post-dose samples in each subject. At these timepoints, the subject will be asked to take the morning dose at the site. Samples collected after 1 week of treatment will be used for the exploratory PK analysis.
Core Phase: Cohort 1 - Change from baseline of the pharmacokinetic (PK) parameter elimination half-life (t1/2) assessed after at least 7 days of dosing. | Baseline up to week 48
  Pharmacokinetic samples will be collected 1 pre-dose in the morning and 3 post-dose (0-2 h, 4-6 h, 6-8 h) after 1 week (Visit 3) and after 6 months (Visit 10). Sampling times will be randomly assigned to each subject to collect at least 1 pre-dose sample and 2 post-dose samples in each subject. At these timepoints, the subject will be asked to take the morning dose at the site. Samples collected after 1 week of treatment will be used for the exploratory PK analysis.
Core Phase: Cohort 2 - Change from baseline of the pharmacokinetic (PK) parameter Area under the concentration-time curve from dosing (time 0) to time t at steady state (AUC0-T,ss). | Baseline up to week 48
  Pharmacokinetic samples will be collected 1 pre-dose in the morning and 3 post-dose (0-2 h, 4-6 h, 6-8 h) after 1 week (Visit 3) and after 6 months (Visit 10). Sampling times will be randomly assigned to each subject to collect at least 1 pre-dose sample and 2 post-dose samples in each subject. At these timepoints, the subject will be asked to take the morning dose at the site. Samples collected after 1 week of treatment will be used for the exploratory PK analysis.
Core Phase: Cohort 2 - Change from baseline of the pharmacokinetic (PK) parameter maximum plasma concentration at steady state (Cmax,ss). | Baseline up to week 48
  Pharmacokinetic samples will be collected 1 pre-dose in the morning and 3 post-dose (0-2 h, 4-6 h, 6-8 h) after 1 week (Visit 3) and after 6 months (Visit 10). Sampling times will be randomly assigned to each subject to collect at least 1 pre-dose sample and 2 post-dose samples in each subject. At these timepoints, the subject will be asked to take the morning dose at the site. Samples collected after 1 week of treatment will be used for the exploratory PK analysis.
Core Phase: Cohort 2 - Change from baseline of the pharmacokinetic (PK) parameter elimination half-life (t1/2) assessed after at least 7 days of dosing | Baseline up to week 48
  Pharmacokinetic samples will be collected 1 pre-dose in the morning and 3 post-dose (0-2 h, 4-6 h, 6-8 h) after 1 week (Visit 3) and after 6 months (Visit 10). Sampling times will be randomly assigned to each subject to collect at least 1 pre-dose sample and 2 post-dose samples in each subject. At these timepoints, the subject will be asked to take the morning dose at the site. Samples collected after 1 week of treatment will be used for the exploratory PK analysis.
Extension Phase: Type, incidence, and severity of treatment-emergent adverse events | postbaseline up to Week 144
Extension Phase: Proportion of patients experiencing treatment-emergent adverse events | postbaseline up to Week 144

SECONDARY OUTCOMES:
Core Phase: Type, incidence, and severity of treatment-emergent adverse events | Baseline up to week 48
Core Phase: Proportion of patients experiencing treatment-emergent adverse events | Baseline up to week 48
Core Phase: Change from baseline as measured by North Star Ambulatory Assessment (NSAA) in cohort 1 after 48 weeks of treatment of givinostat. | Baseline up to week 48
Core Phase: Change from baseline as measured by Bayley III Gross Motor in cohort 2 after 48 weeks of treatment of givinostat. | Baseline up to week 48
Core Phase: Change from baseline in quality of life (as measured by health-related quality of life, HRQOL) at week 48 of treatment of givinostat | Baseline up to week 48

CONTACTS AND LOCATIONS:
Locations (9):
- Queen Fabiola Children's University Hospital HUDERF, Brussels, Belgium
- Italy (3):
  - Fondazione Serena Onlus - Azienda Ospedaliera Niguarda Ca' Granda - NeuroMuscolar Omnicenter, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Policlinico Universitario Agostino Gemelli - Università Cattolica del Sacro Cuore, Roma
- Leids Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- United Kingdom (4):
  - Leeds Teaching Hospital NHS Trust, Leeds, England
  - Great Ormond Street Hospital - GOSH, London, England
  - Newcastle upon Tyne Hospitals NHS Foundation Trust - Newcastle University, Newcastle upon Tyne, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England

IPD SHARING:
Plan to Share IPD: No